CLINICAL TRIAL: NCT06479473
Title: Chemoimmunotherapy Followed by All-residual-lesions Radiotherapy for Extensive-stage Small-cell Lung Cancer: A Phase I/II Trial
Brief Title: Radiotherapy to All Residual Lesions After Chemoimmunotherapy
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Dong Qian, M.D., Anhui Provincial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-ky236
Record Dates: First submitted 2024-06-24; First posted 2024-06-28 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Extensive-stage Small Cell Lung Cancer
Keywords: small-cell lung cancer; extensive-stage; radiotherapy; residual lesion
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Intervention Model Description: All enrolled patients with accordance to the inclusion criteria would first receive 4 to 6 cycles of chemoimmunotherapy (etoposide and cisplatin & carboplatin with Adebrelimab). Then patients who were evaluated as partial response or stable disease would be assigned randomly to receive radiotherapy to all residual lesions followed by Adebrelimab maintenance or only Adebrelimab maintenance up to 2 years.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chemoimmunotherapy group (Active Comparator): Patients assigned to chemoimmunotherapy group would receive 4 to 6 cycles of standard chemoimmunotherapy followed by immunotherapy maintenance to 2 years.
  Interventions: Drug: Chemoimmunotherapy
- Chemoimmunotherapy with radiotherapy group (Experimental): Patients assigned to chemoimmunotherapy group would receive 4 to 6 cycles of standard chemoimmunotherapy followed by radiotherapy to all residual lesions and immunotherapy maintenance to 2 years.
  Interventions: Radiation: Radiotherapy to all residual lesions; Drug: Chemoimmunotherapy

INTERVENTIONS:
Radiation: Radiotherapy to all residual lesions — Patients assigned to chemoimmunotherapy with radiotherapy group would first receive PET-CT and cranial contrasted MRI to ascertain residual lesions. All residual lesions would be irradiated in a hypofractionated manner.
  Arms: Chemoimmunotherapy with radiotherapy group
Drug: Chemoimmunotherapy — atients assigned to chemoimmunotherapy group would receive 4 to 6 cycles of chemoimmunotherapy followed by consolidative immunotherapy

SUMMARY:
Extensive-stage small-cell lung cancer is a lethal malignancy with an extremely poor prognosis. First-line chemotherapy could only achieve an overall survival of approximately 10 months. CREST study demonstrated that the addition of thoracic radiotherapy to the patients who responded to chemotherapy could increase the 2-year survival rate from 3% to 13%. CASPIAN and IMpower 133 trials have established the standard modality of first-line chemoimmunotherapy for extensive-stage small-cell lung cancer and prolonged the overall survival to 13 months. Both the addition of thoracic radiotherapy and immunotherapy to chemotherapy were able to improve the survival. Recently, several retrospective studies have demonstrated the effectiveness and safety of the combination of thoracic radiotherapy and chemoimmunotherapy. In a prospective study, 4-6 cycles of first-line chemotherapy with Adebrelimab followed by thoracic radiotherapy achieved the progression-free survival of 10.1 months and overall survival of 21.4 months, which was longer than chemoimmunotherapy. Another study demonstrated not only thoracic radiotherapy, but also radiotherapy to metastatic lesions could ameliorate survival. Therefore, we supposed that whether radiotherapy to all residual lesions after first-line chemoimmunotherapy could further improve survival for patients with extensive-stage small-cell lung cancer.

DETAILED DESCRIPTION:
Trial design: To enroll 150 patients diagnosed with extensive-stage small-cell lung cancer to receive first-line chemoimmunotherapy with or without radiotherapy to all residual lesions.

Primary endpoint: Progression-free Survival Secondary endpoint: Overall Survival, Objective Response Rate, Duration of Response, Disease Control Rate.

Randomization: All the enrolled patients would be randomly assigned to chemoimmunotherapy group and chemoimmunotherapy with radiotherapy group using random table method.

All enrolled patients with accordance to the inclusion criteria would first receive 4 to 6 cycles of chemoimmunotherapy (etoposide and cisplatin & carboplatin with Adebrelimab). Then patients who were evaluated as partial response or stable disease would be assigned randomly to receive radiotherapy to all residual lesions followed by Adebrelimab maintenance or only Adebrelimab maintenance up to 2 years.

Chemoimmunotherapy: Etoposide 80-100mg/m2 day 1, 2, 3 and cisplatin 75-80mg/m2 day 1 & carboplatin AUC 5 day 1 and Adebrelimab 1200mg day 1 q3w totally 4 to 6 cycles.

Immunotherapy maintenance: Adebrelimab 1200mg q3w to 2 year or disease progression & untolerated toxicity.

Response evaluation: After 4 to 6 cycles of chemoimmunotherapy, patients would undertake response evaluation according to RECIST criteria. These patients who were evaluated as partial response and stable disease could be included into the study and receive randomization.

Radiotherapy to residual lesions: Patients assigned to chemoimmunotherapy with radiotherapy group would first receive PET-CT and cranial contrasted MRI to ascertain residual lesions. All residual lesions would be irradiated in a hypofractionated manner. Radiotherapy should be completed in two weeks. The suggested dose fraction for different lesion was as follows:

Thoracic lesion: 40Gy/10f Cranial lesion: Hippocamps-sparing whole brain irradiation of 30Gy/10f with or without simultaneous integrated lesion boost of 40Gy/10f Hepatic or adrenal lesion: 40Gy/10f Osseous lesion: 30Gy/10f or 40Gy/10f Dose constraint to organs at risk could be referred to QUANTEC criteria (30Gy/10f) and Timmerman's sheet (40Gy/10f) Follow-up: Patients should be follow-up every three months right after the completion of the final cycle of immunotherapy to 3 years after that. Then follow-up every half year is allowed to 5 years. After 5 years, follow-up every year is appropriate. In follow-up, chest CT and abdominal ultrasonography should be implemented. Cranial MRI should be performed every half year. Bone scan should be undertaken every year for all patients.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years old;
* ECOG 0-1;
* Adequate organ function to tolerate chemotherapy, immunotherapy and radiotherapy;
* Small-cell lung cancer;
* Extensive stage confirmed by cranial MRI, chest CT, abdominal ultrasonograph, bone scan or cranial MRI and PET-CT;
* Signature of inform consent.

Exclusion Criteria:

Younger than 18 years old or older than 70 years old;

* ECOG>1;
* Inadequate organ function to tolerate chemotherapy, immunotherapy and radiotherapy;
* Non-small cell lung cancer and other neuroendocrine carcinoma including typical or atypical carcinoid, large-cell neuroendocrine carcinoma;
* Limited stage confirmed by cranial MRI, chest CT, abdominal ultrasonograph, bone scan or cranial MRI and PET-CT;
* No signature of inform consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival | 3 years
  The survival time from diagnose of the disease to progression of the disease

SECONDARY OUTCOMES:
Overall Survival | 3 years
  The survival time from diagnose of the disease to death

CONTACTS AND LOCATIONS:
Overall Officials: Dong Qian, M.D, Principal Investigator — Anhui Provincial Hospital
Locations (1):
- Anhui Provincial Hospital, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No